CLINICAL TRIAL: NCT03103984
Title: Immunosuppression and Diet: the Role of Inflammation in the Adipose Tissue Remodeling After Liver Transplantation
Brief Title: Immunosuppression and Diet: the Role of Inflammation in the Adipose Tissue Remodeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Adaliene Versiani M. Ferreira, PhD, Federal University of Minas Gerais
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 30409114.8.0000.5149
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Liver Transplantation
Keywords: Obesity; Liver transplantation; weight loss diet; immunosuppression
MeSH Terms: conditions — Obesity | interventions — Diet, Reducing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): The volunteers (overweight and obese) will receive nutritional counseling and a weight loss diet.
  Interventions: Other: Weight loss diet
- Immunosuppressed patients (Experimental): The volunteers (liver transplantation) will receive nutritional counseling and a weight loss diet.
  Interventions: Other: Weight loss diet

INTERVENTIONS:
Other: Weight loss diet — Weight loss diet composed of 30% lipids, 30% proteins and 40% carbohydrates.

SUMMARY:
The main goal of this project is to evaluate the effect of immunosuppression in the weight loss and in the metabolic status of patients after liver transplantation. It is also the purpose of this project to investigate why patients become overweight and obese after liver transplantation.

DETAILED DESCRIPTION:
Overweight and obese post-liver transplantation patients will receive a diet to promote weight loss during 6 months. The control group (overweight and obese subjects) will be submitted to the same protocol:

The participants will be interviewed at baseline and after 30, 60, 90 and 180 days from baseline. The following measures will be assessed: body composition (fat body% and free fat body%), anthropometric measures (height, weight, body mass index, waist circumference and abdominal circumference), blood pressure, basal metabolic rate, behavioral symptoms and peripheral biomarkers in the serum. Behavioral symptoms will be assessed using the following self-reported questionnaires: Beck Depression Inventory (depression symptoms), Beck Anxiety Inventory (anxiety symptoms), Medical Outcomes Study 36 - Item Short - Form Health Survey (quality of life) and Perceived Stress Scale (stress).

Enrolled participants will receive a restrictive diet calculated based on individual requirements aiming the loss of around 5%-10% of weight/ 6 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* CONTROL GROUP: Women/men aged 18-60 years old; Body mass index 25-40 kg/m2.
* IMMUNOSSUPPRESSED PATIENTS: Women/men aged 18-60 years old; Body mass index 25-40 kg/m2; liver transplantation between 1-3 years from the time of recruitment.

Exclusion Criteria:

* CONTROL GROUP: Pregnant or lactating womenbuse of alcohol or drugs
* Endocrine disease
* Use of hormones which interferes in the weight
* Use of insulin or anti-inflammatory, and antidepressants drugs
* Use of drugs to loss weight
* Immunosuppressed patients
* Subjects in another weight loss program
* Subjects submitted to bariatric surgery
* IMMUNOSSUPPRESSED PATIENTS: Pregnant or lactating women
* Abuse of alcohol or drugs
* Endocrine disease
* Use of hormones which interferes in the weight
* Use of insulin or antidepressants drugs
* Use of drugs to loss weight
* Subjects in another weight loss program
* Subjects submitted to bariatric surgery, re-transplanted patients, hepatic insufficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in weight measurement from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  The weight loss will be measured by weighing volunteers

SECONDARY OUTCOMES:
Change in body composition from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  The effect of the weight loss diet in body composition will be measured by bioimpedance.
Change in basal metabolic rate from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Basal metabolic rate will be measured by calorimetry.
Change in inflammatory mediators serum levels from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in the levels of interleukins, such as Interleukin-1, interleukin-6 and interleukin-10, interleukin-17, tumor necrosis factor and protein C reactive.
Change in depressive symptoms from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in depressive symptoms will be measured by the Beck Depression Inventory.
Change in anxiety symptoms from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in anxiety symptoms will be measured by the Beck Anxiety Inventory.
Change in quality of life from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in quality of life will be measured by Medical Outcomes Study 36 - Item Short - Form Health Survey.
Change in perceived stress from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in perceived stress will be measured by the Perceived Stress Scale.
Change in quality of diet from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in quality of diet will be measured by the Healthy Eating Index-10.
Changes in serum levels of neurotrophic factors from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in the serum levels of brain-derived neurotrophic factor, glial-derived neurotrophic factor and neurotrophin-3 and neurotrophin 4/5.
Change in metabolic markers serum levels from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Nutritional effect in the levels of triglycerides, cholesterol and glucose
Characterization of the immunological response of liver transplanted patients from baseline until 6 months follow up. | Baseline and 30, 60, 90 and 180 days
  Analysis of cytokines in the sera of immunosupressed patients.
Characterization of the immunological response of liver transplanted patients from baseline until 6 months follow up.. | Baseline and 30, 60, 90 and 180 days
  Analysis of cytokines in cell culture (PBMC) of immunosupressed patients.
Characterization of the immunological profile of liver transplanted patients in the baseline. | Baseline.
  The cells will be immuno-phenotyped for the ex vivo condition and also submitted to culture in the presence of different stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Débora Fernandes Rodrigues, Master, Study Chair — UFMG
Locations (1):
- Hospital da Clínicas da UFMG, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson RA, Garden OJ, Davidson HI. Reduction in energy expenditure after liver transplantation. Nutrition. 2001 Jul-Aug;17(7-8):585-9. doi: 10.1016/s0899-9007(01)00571-8. PMID 11448577
- [Background] Terjimanian MN, Harbaugh CM, Hussain A, Olugbade KO Jr, Waits SA, Wang SC, Sonnenday CJ, Englesbe MJ. Abdominal adiposity, body composition and survival after liver transplantation. Clin Transplant. 2016 Mar;30(3):289-94. doi: 10.1111/ctr.12688. Epub 2016 Feb 13. PMID 26717257
- [Background] Noceti OM, Woillard JB, Boumediene A, Esperon P, Taupin JL, Gerona S, Valverde M, Tourino C, Marquet P. Tacrolimus pharmacodynamics and pharmacogenetics along the calcineurin pathway in human lymphocytes. Clin Chem. 2014 Oct;60(10):1336-45. doi: 10.1373/clinchem.2014.223511. Epub 2014 Aug 20. PMID 25142246
- [Background] Anastacio LR, Diniz KG, Ribeiro HS, Ferreira LG, Lima AS, Correia MI, Vilela EG. Prospective evaluation of metabolic syndrome and its components among long-term liver recipients. Liver Int. 2014 Aug;34(7):1094-101. doi: 10.1111/liv.12495. Epub 2014 Mar 18. PMID 24517561
- [Derived] Rodrigues DF, Fagundes GBP, Monteiro BL, Monteze NM, Rodrigues AMDS, Vieira ELM, Teixeira AL, Teixeira MM, Oliveira MC, Correia MITD, Generoso SV, Ferreira AVM. Blunted inflammatory response is associated with a lower response to a weight loss dietary intervention in liver recipients. Clin Nutr. 2024 Oct;43(10):2438-2447. doi: 10.1016/j.clnu.2024.09.029. Epub 2024 Sep 17. PMID 39305754